CLINICAL TRIAL: NCT00527488
Title: A Single-centre, Open-label, Randomised Explorative Pharmacokinetic/Pharmacodynamic Study of the Gonadotropin-releasing Hormone Receptor Antagonist Degarelix (FE 200486) in Patients With Benign Prostatic Hyperplasia.
Brief Title: Explorative Study of Degarelix for Treatment of Benign Prostatic Hyperplasia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS25; 2007-003578-24 (EudraCT Number)
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2010-11-25 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: BPH
Keywords: Benign Prostate Hyperplasia; BPH; PK/PD; GnRH antagonist
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Degarelix 16+16 mg (Experimental)
  Interventions: Drug: Degarelix
- Degarelix 32 mg (Experimental)
  Interventions: Drug: Degarelix
- Degarelix 32+32 mg (Experimental)
  Interventions: Drug: Degarelix
- Degarelix 64 mg (Experimental)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — Two doses of 16 mg each administered as two administrations (separated by 14 days) will be evaluated for 42 days.
  Arms: Degarelix 16+16 mg
Drug: Degarelix — One dose of 32 mg administered as a single administration will be evaluated for 42 days.
  Arms: Degarelix 32 mg
Drug: Degarelix — Two doses of 32 mg each administered as two administrations (separated by 14 days) will be evaluated for 42 days.
  Arms: Degarelix 32+32 mg
Drug: Degarelix — One dose of 64 mg administered as a single administration will be evaluated for 42 days.
  Arms: Degarelix 64 mg

SUMMARY:
This exploratory study will be conducted open label in a single investigational clinical unit. Altogether 52 patients with benign prostate hyperplasia (BPH) will be randomly assigned to receive 4 different treatments with degarelix.

DETAILED DESCRIPTION:
The present study aims at exploring the potential of the currently available formulation of degarelix to treat BPH with only a short transient lowering of the serum testosterone concentration to or below the castration level defined as 0.5 ng/mL. Two doses and two dosing regimens (32 and 64 mg administered either as a single administration or as two administrations separated by 14 days) will be evaluated for 42 days.

ELIGIBILITY:
Inclusion Criteria:

Each patient must comply with all of the following inclusion criteria to be allowed to be randomised into the study:

1. Man, 55 to 75 years of age.
2. Clinical diagnose of BPH with a prostate volume more than 30 mL, a maximal uroflow of 12 mL/sec or less and an international prostate sympton score (IPSS) of 13 or more at screening.
3. A prostate specific antigen (PSA) value less than 10 ng/mL and no clinical evidence of adenocarcinoma of the prostate at screening. If a biopsy of the prostate is performed, a period of 6 weeks should be allowed after the biopsy before the patient is enrolled into the study.
4. Has a baseline testosterone level above 3 ng/mL at screening.

Exclusion Criteria:

Any patient meeting one or more of the following exclusion criteria will not be included into the study:

1. Previous surgery of the prostate.
2. Previous treatment with GnRH agonists or GnRH antagonists.
3. Treatment with 5-alpha reductase inhibitors, e.g., finasteride (Prosca®)or dutasteride (Avodart®) within the past 12 months before the study.
4. Treatment with alpha-adrenergic antagonists, e.g., terazosin, doxazosin, tamsulosin, alfuzosin within 2 weeks prior to Screening part II (or Part I, if IPSS is performed at Screening part I).
5. Treatment with any drug modifying the testosterone level or function within 12 weeks before Screening visit part II (or Part I, if IPSS is performed at Screening part I).

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- CRS Clinical Research Services Monchengladback GmbH, Mönchengladbach, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Degarelix 16+16 mg: Two doses of Degarelix 16 mg on Day 0 and Day 14
- Degarelix 32 mg: A single dose of Degarelix 32 mg on Day 0
- Degarelix 32+32 mg: Two doses of Degarelix 32 mg on Day 0 and Day 14
- Degarelix 64 mg: A single dose of Degarelix 64 mg on Day 0
Period: Overall Study
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Started | 13 | 13 | 13 | 13
Completed | 13 | 12 | 12 | 13
Not Completed | 0 | 1 | 1 | 0
Not completed — Withdrawn prior to dosing | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg | Total
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (4.7) | 63.0 (6.1) | 66.3 (4.6) | 60.4 (7.8) | 63.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 13 | 13 | 13 | 13 | 52
Region of Enrollment [Number; unit: participants]
  Germany | 13 | 13 | 13 | 13 | 52

OUTCOME MEASURES:

1. Primary Outcome: Testosterone Area Below Baseline Interval
Description: The area of the testosterone concentration (ng/mL) vs. time (days) curve that is below the baseline interval concentration( i.e. 0.75 x baseline concentration)
Time Frame: 0-42 Days
Measure: Mean (Standard Deviation); unit: ng*days/mL
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
ng*days/mL | 21.0 (19.1) | 16.0 (11.6) | 54.6 (25.7) | 70.6 (53.9)

2. Secondary Outcome: Pharmacokinetic Parameters of Degarelix: AUCt
Description: Area under the time-concentration curve (AUCt) was calculated by non-compartmental methods based on data up to Day 42
Time Frame: 0-42 Days
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
ng*day/mL | 70.7 (20.6) | 86.9 (26.9) | 158 (43.7) | 176 (47.2)

3. Primary Outcome: Time of Testosterone Concentration Below Baseline Interval
Description: The time from when the testosterone concentration falls below the baseline interval limit (i.e. 0.75 x baseline concentration) until it returns above this limit
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
Days | 21.2 (12.8) | 13.2 (9.3) | 34.3 (10.8) | 34.0 (11.7)

4. Primary Outcome: Minimal Value of Testosterone (Cnadir)
Description: The lowest concentration of testosterone measured within the time frame
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
ng/mL | 1.4 (0.5) | 0.9 (0.5) | 0.4 (0.3) | 0.4 (0.2)

5. Primary Outcome: Time of Minimal Value of Testosterone (Tnadir)
Description: The time point when the lowest testosterone concentration was measured
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
Days | 1.1 (0.6) | 1.3 (0.8) | 4.3 (5.3) | 8.8 (9.9)

6. Primary Outcome: Duration of Testosterone Concentration Below 0.5 ng/mL
Description: The time from when the testosterone concentration falls below 0.5 ng/mL until it returns above that level
Time Frame: Day 0-42
Measure: Median (Full Range); unit: Days
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
Days | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 2.2] | 1.4 [0.0 to 41.1] | 2.0 [0.0 to 41.1]

7. Primary Outcome: Number of Subjects With Testosterone Concentration ≤0.5 ng/mL
Time Frame: Day 0-42
Measure: Number; unit: participants
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
participants
  Day 1 | 0 | 2 | 5 | 8
  Day 5 | 0 | 0 | 1 | 2
  Day 14 | 0 | 0 | 1 | 5
  Day 17 | 0 | 0 | 8 | 5
  Day 28 | 0 | 0 | 3 | 5
  Day 42 | 0 | 0 | 3 | 5

8. Primary Outcome: Number of Subjects With Testosterone Concentration at or Above the Baseline Interval Concentration
Description: The baseline interval concentration is 0.75 x baseline concentration
Time Frame: Day 0-42
Measure: Number; unit: participants
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
participants
  Day 1 | 0 | 0 | 0 | 0
  Day14 | 11 | 10 | 7 | 2
  Day 28 | 8 | 9 | 3 | 3
  Day 42 | 8 | 12 | 3 | 4

9. Primary Outcome: Prostate Specific Antigen (PSA) Concentration
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
ng/mL
  Baseline | 3.9 (3.2) | 3.0 (2.6) | 2.8 (2.5) | 3.2 (3.1)
  Day 42 | 3.7 (2.5) | 2.5 (1.7) | 2.4 (2.6) | 2.3 (1.9)

10. Primary Outcome: Prostate Volume
Description: The prostatic volume was measured by transrectal ultrasound. The prostatic gland was sonicated from two directions perpendicular to one another resulting in three cursor positions set by the urologist, and the volume automatically calculated.
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
mL
  Baseline | 42.0 (12.1) | 48.7 (21.0) | 38.1 (7.1) | 38.9 (9.0)
  Day 42 | 34.5 (11.0) | 34.8 (14.2) | 28.7 (8.2) | 30.6 (10.5)

11. Primary Outcome: Maximal Urinary Flow
Description: Urinary flow was determined by flowmetry using a device that fulfils the International Continence Society standards for maximum urinary flow.
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
mL/s
  Baseline | 10.0 (4.7) | 11.7 (3.4) | 9.7 (4.1) | 9.1 (3.0)
  Day 42 | 10.1 (4.3) | 11.2 (4.0) | 12.2 (9.3) | 11.9 (9.1)

12. Primary Outcome: Post-void Residual Urine Volume
Description: The post-void residual urine volume in the bladder was evaluated by transabdominal ultrasound. The urine bladder was sonicated from two directions perpendicular to one another, and the volume calculated automatically.
Time Frame: Day 0-42
Measure: Mean (Full Range); unit: mL
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
mL
  Baseline | 63.4 [4.8 to 170] | 60.7 [0.0 to 157] | 56.7 [8.4 to 201] | 91.3 [4.6 to 368]
  Day 42 | 58.0 [0.3 to 215] | 45.2 [0.0 to 108] | 34.6 [0.0 to 165] | 75.8 [0.0 to 259]

13. Primary Outcome: International Prostate Specific Symptom (IPSS) Score
Description: The IPSS is a patient-administered questionnaire containing seven items to evaluate symptoms of urinary obstruction (incomplete emptying, frequency, hesitancy, urgency, weak stream, straining, nocturia) over the preceding week. Each urinary symptom question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (0-7: mildly symptomatic; 8-19: moderately symptomatic; 20-35: severely symptomatic).
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
Units on a scale
  Baseline | 17.7 (4.5) | 22.3 (6.5) | 18.2 (5.4) | 21.8 (6.2)
  Day 42 | 11.6 (4.5) | 9.1 (6.2) | 8.6 (5.7) | 11.8 (5.9)

14. Primary Outcome: IPSS Global Quality of Life
Description: Patients were asked about how they would feel if they were to spend the rest of their lives with their prostate symptoms just as they are now. The answers choices range from "delighted" to "terrible" or 0 to 6.
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
Units on a scale
  Baseline | 4.2 (1.1) | 3.8 (1.7) | 4.3 (1.3) | 4.7 (1.4)
  Day 42 | 2.9 (1.4) | 1.8 (2.0) | 1.9 (1.6) | 2.5 (1.3)

15. Primary Outcome: Interntional Iindes of Erectile Function (IIEF) Score: Overall Satisfaction
Description: The IIEF contains 15 items in 5 domains: Erectile Function (6 items), Orgasmic Function (2 items), Sexual Desire (2 items), Intercourse Satisfaction (3 items), and Overall Satisfaction (2 items). Item are scored on a scale from 'No sexual activity' to 'Almost always to always'. For the Erectile Function domain, a score of 1-10 indicates severe erectile dysfunction and 26-30 no dysfunction, the minimum score being 1 and the maximum 30. For all other domains, a higher score indicates less dysfunction. The IIEF does not yield a total score.
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
Units on a scale
  Baseline | 6.6 (1.8) | 6.5 (2.5) | 5.8 (2.6) | 5.9 (2.8)
  Day 42 | 6.8 (1.8) | 6.2 (3.2) | 6.0 (3.0) | 5.1 (2.3)

16. Secondary Outcome: Pharmacokinetic Parameters of Degarelix: Cmax
Description: Cmax was determined for concentration measurements up to Day 42
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
ng/mL | 4.5 (1.2) | 6.9 (1.9) | 9.6 (3.0) | 15.8 (4.6)

17. Secondary Outcome: Pharmacokinetic Parameters of Degarelix: Tmax
Description: The time for maximal concentration (tmax) was determined for data up to Day 42
Time Frame: Day 0-42
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Number analyzed (Participants) | 13 | 12 | 12 | 13
Days | 1.0 (0.0) | 1.3 (0.8) | 1.1 (0.6) | 1.1 (0.6)

ADVERSE EVENTS:
Time Frame: Day 0-42
Arm/Group | Degarelix 16+16 mg | Degarelix 32 mg | Degarelix 32+32 mg | Degarelix 64 mg
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 1/12 | 1/13
Other Adverse Events (participants affected / at risk) | 13/13 | 11/12 | 12/12 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 16+16 mg (N=13) | Degarelix 32 mg (N=12) | Degarelix 32+32 mg (N=12) | Degarelix 64 mg (N=13)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Causality to degarelix regarded as unlikely by the investigator
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Causality regarded as unlikely by the investigator
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 16+16 mg (N=13) | Degarelix 32 mg (N=12) | Degarelix 32+32 mg (N=12) | Degarelix 64 mg (N=13)
Injection site reaction (Injury, poisoning and procedural complications) | 11 (29) | 11 (25) | 12 (39) | 13 (37)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of libido (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Libido increased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the end of the study, one or more manuscripts for joint publication may be prepared in collaboration between the investigator(s) offered authorship and Ferring Pharmaceuticals A/S (Ferring). Ferring reserves the right to be last author(s) in all publications related to this study. In the event of any disagreement in the content of any publication, both the Investigator's and Ferring's opinion will be fairly and sufficiently represented in the publication.